CLINICAL TRIAL: NCT03612921
Title: Oral Amantadine Versus IV Amantadine to Attenuate the Hemodynamic Response to Laryngoscopy, Tracheal Intubation and Surgical Incision and Their Effect on β-endorphin: A Randomized Clinical Trial
Brief Title: Oral Amantadine, IV Amantadine and Hemodynamic Response to Laryngoscopy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ghada Mohammed AboelFadl, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 17300205
Record Dates: First submitted 2018-05-16; First posted 2018-08-02 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Intubation, Intratracheal
Keywords: oral amantadine; IV amantadine; tracheal intubation
MeSH Terms: interventions — Amantadine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind (Subject, Caregiver, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- oral group (Active Comparator): the patients will receive oral amantadine sulfate using the dose 100 mg 90 minute prior to the surgery and infusion of100cm I.V saline
  Interventions: Drug: oral Amantadine sulfate
- I.V group (Active Comparator): the patients will receive 100 mg I.V amantadine sulfate infusion over 60minute prior to the surgery and placebo tablet 90 minute prior to the surgery
  Interventions: Drug: i.v Amantadine Sulfate
- control group (group C) (Placebo Comparator): the patients will receive placebo tablet 90 minute prior to the surgery and infusion of 100cm I.V saline over 60minute prior to the surgery
  Interventions: Drug: placebo tablet

INTERVENTIONS:
Drug: oral Amantadine sulfate — oral amantadine
  Other Names: amantadine
  Arms: oral group
Drug: i.v Amantadine Sulfate — intra venous amantadine
  Other Names: PK-Merz
  Arms: I.V group
Drug: placebo tablet — placebo tablet
  Arms: control group (group C)

SUMMARY:
this study will be undertaken-to evaluate the effect of oral amantadine versus IV amantadine premedication on the hemodynamic response to laryngoscopy ,tracheal intubation and surgical incision and their effect on β-endorphins.

DETAILED DESCRIPTION:
Direct laryngoscopy and passage of endotracheal tube through the larynx is a noxious stimulus, which can provoke untoward response in the cardiovascular, respiratory and other physiological systems .Amantadine is a non-competitive NMDA receptor antagonist, and compared to ketamine, it is well tolerated with fewer side effects (mainly dizziness, sedation, and dry mouth). Amantadine's formulation permits the oral route for drug delivery, as well as the IV route. The side-effects profile of amantadine via all routes seems not to be harmful in appropriate dosages.. Amantadine has been clinically used as an antiviral drug, for dementia, and in the treatment of Parkinson's disease and spasticity. It is a non-competitive NMDA receptor antagonist, and compared to ketamine, it is well tolerated with fewer side effects (mainly dizziness, sedation, and dry mouth). Amantadine's formulation permits the oral route for drug delivery, as well as the IV route. The side-effects profile of amantadine via all routes seems not to be harmful in appropriate dosages.

In the central nervous system, beta-endorphins bind mu-opioid receptors and exert their primary action at presynaptic nerve terminals. However, instead of inhibiting substance P, they exert their analgesic effect by inhibiting the release of GABA, an inhibitory neurotransmitter, resulting in excess production of dopamine.

this study will be undertaken-to evaluate the effect of oral amantadine versus IV amantadine premedication on the hemodynamic response to laryngoscopy ,tracheal intubation and surgical incision and their effect on β-endorphins.

ELIGIBILITY:
Inclusion Criteria:

* ASA I&II
* the age range 20-55 years scheduled for elective back surgery(laminectomy, discectomy and spinal canal stenosis)

Exclusion Criteria:

* Patient refusal
* Patients with ASA score III (with chronic kidney, lungs, Gastrointestinal tract, liver, or cardiovascular diseases)
* Pregnant or breastfeeding women.
* Allergy to any of the study medications and taking medications that could significantly interact with amantadine (tramadol, atropine, antipsychotic medications)
* DM, thyroid disease any endocrine disease
* Suspected difficult intubation or intubation time more than 30 second.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-08-15 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
the effect of oral amantadine versus IV amantadine premedication on laryngoscopy and tracheal intubation on β-endorphins . | baseline( before medication) , 5 minutes before induction of anaesthesia, 3 minutes after induction , 5 minutes after tracheal intubation and 5 minutes after skin incision
  changes of the mean arterial blood pressure (mmhg)

SECONDARY OUTCOMES:
the effect of oral amantadine versus IV amantadine premedication on the hemodynamic response to surgical incision | 2 blood samples one just before medication and the second after 10 minutes after skin incision
  β-endorphins level in the blood

CONTACTS AND LOCATIONS:
Overall Officials: Ghada Abu El Fadl, MD, Principal Investigator — Assiut, Assiut governorate, Egypt, 715715
Locations (1):
- Assiut university hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided